CLINICAL TRIAL: NCT05613244
Title: Orbital Solitary Fibrous Tumors: Description of a Case Series and Study of the Recurrence Rate
Brief Title: Descriptive Study of a Cohort of Orbital Solitary Fibrous Tumors
Acronym: TFS-ORB
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NMR_2020_36
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Orbital Tumor
MeSH Terms: conditions — Orbital Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Orbital Solitary Fibrous Tumors
  Interventions: Other: Phone call

INTERVENTIONS:
Other: Phone call — Patients will be asked to complete a questionnaire via a phone call

SUMMARY:
Orbital solitary fibrous tumors are rare tumors with an intermediate potential of malignancy. Orbital solitary fibrous tumors' prognostic criteria are still poorly understood.

Some patients with orbital solitary fibrous tumors have been treated at the Adolphe de Rothschild Foundation Hospital. This cohort will be studied to describe the recurrence rate and to identify predictive factors of recurrence or metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at the Adolphe de Rothschild foundation hospital for an orbital solitary fibrous tumor between 01/01/2014 and 09/30/2020

Exclusion Criteria:

* Opposition of the patient (or of the relative if the patient is deceased)
* Patients benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an orbital solitary fibrous tumor
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Population characteristics | inclusion
  descriptive statistics of each variable: age, sex, symptoms, duration of symptoms
Medical history | inclusion
  descriptive statistics of each variable: history of previous biopsy or excision, previous intraoperative data,previous pathological data
Radiological lesion features | inclusion
  descriptive statistics of each variable: laterality, orbital location, size and characteristics on preoperative orbital imaging
Pathological lesion characteristics | inclusion
  descriptive statistics of each variable: presence of necrosis, presence of epithelioid morphology of these cells, presence of cellular atypia, description of the mitotic index, immunohistochemical study, proliferation factor
Intraoperative data | inclusion
  descriptive statistics of each variable: complete or incomplete surgical removal, surgical removal 'in toto' or by fragments

CONTACTS AND LOCATIONS:
Overall Officials: Natasha MAMBOUR, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France